CLINICAL TRIAL: NCT01271673
Title: A Short Duration Pilot Cohort Study to Assess the Level of Compliance in Undertaking Breast Self Examination (BSE) Among Women Attending Preventive Oncology Clinic
Brief Title: Cohort Study to Assess the Level of Compliance in Undertaking Breast Self Examination Among Women Attending Preventive Oncology Clinic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Tata Memorial Hospital, Tata Memorial Hospital
Other Study IDs: 827
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-11

CONDITIONS: Breast Self Examination
MeSH Terms: conditions — Breast Self-Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Women undertaking Breast Self Examination: Women attending Preventive Oncology Clinic during the month of November- December 2010,and undertaking BSE training whose Residential address mentioned as Mumbai and whose Contact number is available.

SUMMARY:
Breast cancer is the most common cancer among women residing in majority of the urban areas in India. The deaths due to breast cancer are mainly a result of late presentation of the symptoms due to lack of awareness of the signs and symptoms of the disease and lack of knowledge of performing BSE. The BSE technique can be a good tool for improving the awareness about the symptoms of breast cancer. Hence, we propose a pilot study of short duration (3 months follow-up), to assess the level of compliance to BSE and assess the various reasons for non-compliance. Based on the results of this study a long term cohort study will be planned with similar objectives.

DETAILED DESCRIPTION:
This is an observational cohort study about BSE among women attending the Preventive Oncology (PO) Clinic, TMH. All women attending for screening of common cancers at the Preventive Oncology OPD at TMH are demonstrated the technique of BSE and advised on when, how and why to perform BSE.

Women attending the PO clinic and who have mentioned their residential address as Mumbai and provided contact number will be invited to participate in the study. They will be explained the study protocol and those who are interested in participating will be offered informed consent forms. The women who sign the informed consent form will be enrolled into the trial.

The data regarding the socio-demographic details and level of knowledge, attitude and practice (KAP) about breast cancer and BSE will be collected from the participating women. They will be asked if they have any doubts regarding the technique of BSE and their willingness to perform BSE. Thereafter, a follow-up period of 3 months, the women will be contacted telephonically to collect the data to assess the level of compliance to BSE and the reasons for non-compliance, if any. Also, the compliant women will be asked if they have observed any abnormal changes in their breasts and have they visited the clinician for the same. And subsequently, their health care seeking behaviour will be studied.

The data collected before and after the follow-up will be entered in the SPSS software and analyzed using simple statistical tests like mean, chi-square, t-test and univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women attending Preventive Oncology Clinic during the month of November-December 2010.
* Women undertaking BSE training.
* Residential address mentioned as Mumbai.
* Contact number available.

Exclusion Criteria:

* Women residing outside Mumbai, Maharashtra.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women attending Preventive Oncology Clinic in the month of November-December 2010.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Compliance to Breast Self Examination | 3 months
  To assess the level of compliance in undertaking Breast Self Examination among women attending Preventive Oncology Clinic.

SECONDARY OUTCOMES:
Association of various socio-demographic factors and the level of compliance to Breast Self Examination | 3 months
  To study the association of various socio-demographic factors and level of compliance with Breast Self Examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ketaki G Karnik, MSc, Principal Investigator — University of Pune; Gauravi A Mishra, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Department of Preventive Oncology, Tata Memorial Hospital, Mumbai, Maharashtra, India